CLINICAL TRIAL: NCT05664438
Title: Multimodal MRI to Differentiate Subtypes of Intramedullary Spinal Cord Tumours: A Pilot Study
Brief Title: 3T MRI of Intramedullary Spinal Cord Tumours
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 15346
Record Dates: First submitted 2022-12-05; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Spinal Cord Tumor of Cervical Spine
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI scan — MRI scan of cervical spine

SUMMARY:
Intramedullary spinal cord tumours (IMSCTs) are a type of tumour that arises from cells within the spinal cord. They are rare, accounting for around 4-10% of central nervous system tumours. They commonly present as back/neck pain and have poor outcomes if not treated.

IMSCTs fall into various subtypes. Around 90% are either ependymomas or astrocytomas. Ependymomas are usually quite distinct from the surrounding tissue and therefore can often be treated successfully with surgery. In contrast, astrocytomas tend to invade the surrounding tissue and, as a result, generally cannot be entirely surgically removed. Radiotherapy is recommended instead of surgery for tumours that cannot be operated. Unfortunately, ependymomas and astrocytomas can appear very similar on diagnostic scans and are therefore difficult to tell apart before surgery. Biopsy therefore remains the current gold standard for tumour subtype differentiation.

Any spinal cord surgery, whether it be biopsy or resection, poses major challenges due to the small size of the spinal cord. A small corridor via the back of the spinal cord, known as the posterior midline, usually offers the safest approach to a tumour. However, finding this access corridor can be very difficult because tumours tend to deform the anatomy of the spinal cord, leading to a high risk of injury to the normal spinal cord tissue or nerves.

The primary objective of this pilot study is to test if cutting-edge spinal cord magnetic resonance imaging (MRI) techniques could help to better differentiate between tumour subtypes. The investigators will do this by comparing various imaging metrics between the tumour subtypes, confirmed by biopsy. The investigators' second objective is to see if these MRI techniques could help to identify, pre-surgery, the location of the posterior midline of the spinal cord. The investigators will do this by comparing the prediction of the midline location from imaging with blinded observations by the surgeon during planned surgery. Additionally, the investigators want to investigate the relationship between imaging metrics and patient pain and sensorimotor symptoms, to explore if imaging offers insight into the variety of clinical symptoms associated with these tumours.

The investigators' hope is that the results of this study could inform a future larger trial that would be designed to fully assess the utility of cutting-edge MRI techniques for reducing both the need for spinal cord surgery and the risks associated with surgery in IMSCT patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above
* Radiological diagnosis of IMSCT in the cervical spinal cord
* Planned to undergo a biopsy or has already undergone a biopsy to determine tumour subtype
* Sufficient remnant tumour as decided by the study team by review of patients clinical radiological scans

Exclusion Criteria:

* Contraindication to MRI, including certain metal implants
* Subjects who are pregnant or planning pregnancy
* Any previous therapy that could in the opinion of the CI confound the research MRI characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be patients with a diagnosis of IMSCT in the cervical region of the spinal cord. We will aim to recruit approximately 50% ependymoma and 50% astrocytoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether advanced MRI can differentiate between tumour subtypes confirmed by histopathology from biopsy | Study visit
  Compare structural MR imaging metrics, metabolic MR imaging metrics and clinical radiology evidence of bone remodelling, presence of syrinx and presence of haemorrhage between tumour subtypes.

SECONDARY OUTCOMES:
Determine the added value of advanced MRI features to identify the spinal cord posterior midline | Study visit and surgery
  Compare variations in tissue signal intensity, asymmetry in Tract Density Imaging and asymmetry in vasculature with surgical metrics.
Investigate the relationship between MRI metrics and patient pain and sensorimotor symptoms | Study visit and surgery
  Compare functional MRI activity, functional MRI connectivity and tumour volume/location with pain scores, pain questionnaires, sensorimotor questionnaires/diagrams, overall function scores and overall function questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No